CLINICAL TRIAL: NCT01304992
Title: Effects of Lupin Protein on Lipid and Protein Metabolism in Moderate Hypercholesterolemic Subjects
Brief Title: Cholesterol-lowering Effects of Lupin Protein
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: German Federal Ministry of Education and Research (Other Government)
Responsible Party: Principal Investigator, Gerhard Jahreis, Prof. Dr. habil., University of Jena
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: LSEP H48-11
Record Dates: First submitted 2011-02-25; First posted 2011-02-28 (Estimated); Last update posted 2012-11-27 (Estimated); Status verified 2012-11

CONDITIONS: Hypercholesterolemia
Keywords: Dietary protein; Lupin protein; Cholesterol metabolism; Protein metabolism; Hypercholesterolemia; Protein-enriched drinks
MeSH Terms: conditions — Hypercholesterolemia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Lupin Protein (Experimental): Lupin protein (cultivar: Lupinus angustifolius Boregine; incorporated in a drink)
  Interventions: Dietary Supplement: Protein drink - low dosage; Dietary Supplement: Protein drink - high dosage
- Reference protein (Active Comparator): Reference Protein (75% sodium caseinate (EM7; DMV international) and 25% milk protein (Megglosat HP; Meggle), incorporated in a drink)
  Interventions: Dietary Supplement: Protein drink - low dosage; Dietary Supplement: Protein drink - high dosage
- Wash out (No Intervention): Wash out (four weeks without any intervention between interventional periods)

INTERVENTIONS:
Dietary Supplement: Protein drink - low dosage — The subjects will consume 500 mL of a protein drink containing 25 g protein (lupin protein or reference protein) per day over eight weeks each. After a one-week run-in period, each volunteer has to pass both protein-periods in different order with a four-week wash out period in between.
  Arms: Lupin Protein; Reference protein
Dietary Supplement: Protein drink - high dosage — The subjects will consume 500 mL of a protein drink containing 40 g protein (lupin protein or reference protein) per day over eight weeks each. After a one-week run-in period, each volunteer has to pass both protein-periods in different order with a four-week wash out period in between.
  Arms: Lupin Protein; Reference protein

SUMMARY:
The objective of the study is to determine the efficacy of lupin protein drinks (Lupinus angustifolius Boregine) in humans. Parameters concerning cardiovascular risk factors and the metabolism of proteins, lipids and cholesterol will be evaluated.

DETAILED DESCRIPTION:
Based on the preliminary finding that a daily dosage of 35 g lupin protein is capable to affect plasma lipids positively, the physiological effects of two different daily lupin protein dosages will be investigated in two separate study groups (group A: 25 g protein/day; group B: 40 g protein/day). Both study groups undergo double-blinded and controlled study conditions in a cross-over design.

In each of the two study groups 35 volunteers with hypercholesterolemia will be allocated to one of two randomization groups: After a 1-week run-in period (baseline), half of the 35 participants of each study group will consume drinks with lupin protein in the respective amount (25 g or 40 g protein/day) over a period of eight weeks, the other half will receive the analogue amount of milk protein as well incorporated in a drink serving as control. After a wash-out period of four weeks, the protein source will be crossed within the two study groups for a second intervention period of eight weeks.

ELIGIBILITY:
Inclusion Criteria:

* Moderate hypercholesterolemia (total cholesterol >5,2 mmol/L)
* Age: 18-80 years old

Exclusion Criteria:

* Intake of lipid-lowering pharmaceuticals
* Allergy against legumes or milk protein
* Intolerance against milk
* Pregnancy, lactation
* Chronic bowel disease

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 66 (Actual)
Dates: Start 2011-02; Primary Completion 2011-08 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Cholesterol metabolism | After 0, 4, 8, 12, 16 and 20 weeks
  Blood lipids (LDL cholesterol, total cholesterol, HDL cholesterol, triacylglyceroles)

SECONDARY OUTCOMES:
Protein metabolism | After 0, 8, 12 and 20 weeks
  Plasma: amino acids, total protein, albumin, urea, uric acid; Urine: total protein, ammonia, urea, uric acid; Proteomic-study
Body composition (body status) | After 0, 8, 12 and 20 weeks
  Bioelectrical impedance analysis, body weight, blood pressure
High-sensitive CRP | After 0, 8, 12 and 20 weeks
  As inflammation marker
Fasting glucose | After 0, 8, 12 and 20 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Gerhard Jahreis, Prof. Dr., Principal Investigator — Friedrich Schiller University Jena, Institute of Nutrition, Department of Nutritional Physiology
Locations (1):
- Friedrich Schiller University Jena, Department of Nutritional Physiology, Jena, Thuringia, Germany

REFERENCES:
- [Derived] Bahr M, Fechner A, Kramer J, Kiehntopf M, Jahreis G. Lupin protein positively affects plasma LDL cholesterol and LDL:HDL cholesterol ratio in hypercholesterolemic adults after four weeks of supplementation: a randomized, controlled crossover study. Nutr J. 2013 Aug 1;12:107. doi: 10.1186/1475-2891-12-107. PMID 23902673